CLINICAL TRIAL: NCT02384629
Title: PCI With AXXESS Biolimus A9 Eluting Bifurcation Stent in Treating Coronary Artery Bifurcation Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Problem with medical device provider
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2014-0079
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Bifurcation Lesions
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AXXESS stent1 (Experimental): AXXESS stent (OCT-guided)
  Interventions: Device: OCT-guided PCI with AXXESS stent
- Conventional DES1 (Experimental): Conventional DES (Biomatrix flex stent, OCT-guided)
  Interventions: Device: OCT-guided PCI with conventional DES (Biomatrix flex stent)
- AXXESS stent2 (Active Comparator): AXXESS stent (Angio-guided)
  Interventions: Device: Angio-guided PCI with AXXESS stent
- Conventional DES2 (Active Comparator): Conventional DES (Biomatrix flex stent, Angio-guided)
  Interventions: Device: Angio-guided PCI with PCI with conventional DES (Biomatrix flex stent)

INTERVENTIONS:
Device: OCT-guided PCI with AXXESS stent — The AXXESS stent (Biosensors Europe SA, Morges, Switzerland) is a dedicated self-expanding bifurcation stent eluting the sirolimus analog Biolimus A9 emulsed in a biodegradable polymer. It has the advantage to preserve the ostium of both distal branches and allows additional stent implantation in the distal branches for complete lesion coverage, while reducing large stent overlap and eliminating deformation. Optical coherence tomography (OCT), has enabled the evaluation of strut coverage and arterial healing after DES implantation with a superior resolution and delineation over other imaging modalities. With using these superiorities of OCT, there have been many studies assessing the neointimal coverage following various types of DES implantation in various periods.
  Arms: AXXESS stent1
Device: OCT-guided PCI with conventional DES (Biomatrix flex stent) — BioMatrix Flex is abluminal biodegradable polymer DES. Its abluminal coating is absorbed after 6 to 9months and turns the DES into a BMS. It combines the proven safety of a DES with an abluminal biodegradable polymer, the prove efficacy of BA9 and an advanced stent design. Optical coherence tomography (OCT), has enabled the evaluation of strut coverage and arterial healing after DES implantation with a superior resolution and delineation over other imaging modalities. With using these superiorities of OCT, there have been many studies assessing the neointimal coverage following various types of DES implantation in various periods.
  Arms: Conventional DES1
Device: Angio-guided PCI with AXXESS stent — The AXXESS stent (Biosensors Europe SA, Morges, Switzerland) is a dedicated self-expanding bifurcation stent eluting the sirolimus analog Biolimus A9 emulsed in a biodegradable polymer. It has the advantage to preserve the ostium of both distal branches and allows additional stent implantation in the distal branches for complete lesion coverage, while reducing large stent overlap and eliminating deformation. We use the conventional coronary angiography.
  Arms: AXXESS stent2
Device: Angio-guided PCI with PCI with conventional DES (Biomatrix flex stent) — BioMatrix Flex is abluminal biodegradable polymer DES. Its abluminal coating is absorbed after 6 to 9months and turns the DES into a BMS. It combines the proven safety of a DES with an abluminal biodegradable polymer, the prove efficacy of BA9 and an advanced stent design. We use the conventional coronary angiography.
  Arms: Conventional DES2

SUMMARY:
1. To compare the safety and efficacy of AXXESS stent with conventional DES in patients with coronary artery bifurcation disease
2. To assess the impact of optical coherence tomography (OCT) guidance on clinical outcomes following the stent type

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures,
* Patients ≥ 19 years old,
* Patients who are expected to undergo PCI for bifurcation lesions.

Exclusion Criteria:

* Age> 85 years,
* Cardiogenic shock or unstable patients,
* Increased risk of bleeding, anemia, thrombocytopenia,
* A need for oral anticoagulation therapy,
* Pregnant women or women with potential childbearing,
* Life expectancy < 1 year.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Late loss of side branch(SB) | 9 months after procedure
  Late loss was defined as the difference between the minimal luminal diameter (MLD) immediately after the procedure and the MLD at 9-month follow-up, Measured the change in MLD by Quantitative coronary angiography (QCA)

SECONDARY OUTCOMES:
Cardiovascular (CV) death | 9 months after procedure
  death for CV cause (MI, stroke)
Myocardial infarction (MI) | 9 months after procedure
  MI definition: rise of cardiac biomarker with at least one of the following: Symptoms of ischemia, New or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB), Development of pathological Q waves in the ECG, Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality, identification of an intracoronary thrombus by angiography or autopsy
stent thrombosis (ST) | 9 months after procedure
  ST definition: Academic Research Consortium (ARC) definition
SB closure | 9 months after procedure
  SB closure: TIMI flow < 3 and/or stenosis >75%